CLINICAL TRIAL: NCT02538133
Title: Tomoscintigraphie Hybride Aux Leucocytes Marqués Dans le Diagnostic Des Infections de Prothèses Vasculaires.
Brief Title: Study Assessing Hybrid SPECT-CT With Labeled Leukocytes for Diagnosis of Vascular Prosthesis Infections
Acronym: LEUCOPRO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 49RC14_0072; 2015-001342-28 (EudraCT Number)
Record Dates: First submitted 2015-07-30; First posted 2015-09-02 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2015-08

CONDITIONS: Vascular Prosthesis Infection
Keywords: 99mTc-Exametazime (HMPAO)-Labeled Leukocytes; suspected subdiaphragmatic vascular prosthesis infection; diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 99mTc-Exametazime (HMPAO)-labeled leucocytes (Experimental)
  Interventions: Biological: 99mTc-Exametazime (HMPAO)-labeled leukocytes

INTERVENTIONS:
Biological: 99mTc-Exametazime (HMPAO)-labeled leukocytes — Hybrid tomoscintigraphy with labeled leucocytes for patients with suspected vascular prosthesis infection

SUMMARY:
Vascular Prothesis Infection is a rare but an extremely serious complication. Diagnosis is often difficult (germs are found only in 50% of cases). Conventional imagery is often non-specific and difficult to interpret especially in early postoperative phase. Leukocytes isolated from the patient's blood are labeled with a radiopharmaceutical technetium 99mTc-HMPAO.

The aim of this study is to assess the overall diagnostic performance of scintigraphy (hybrid SPEC-CT) with labeled leucocytes in diagnosis of subdiaphragmatic vascular prothesis infection.

ELIGIBILITY:
Inclusion Criteria:

* patient of more than 18 years old
* Patient with a subdiaphragmatic vascular prosthesis
* Vascular prosthesis infection suspected with clinical (flow from the scare and/or local pain and/or erythema and/or persistent fever and/or bacteraemia) and/or biological (inflammatory syndrome : elevated C-reactive protein and/or erythrocyte sedimentation rate (ESR) and/or white blood cells increased) infection signs
* Patient willing to participate with a signed informed consent
* Patient covered by a healthcare insurance

Exclusion Criteria:

* Pregnant women or of childbearing age without effective contraception
* Prosthesis limited to a bare stent.
* Patient who has been committed to an institution by legal or regulatory order
* Contraindications for labeled leukocytes scintigraphy realization :
* Restlessness, inability to keep still lie at least 1 hour
* Claustrophobia
* Poor compliance predictable or impaired general condition making it impossible to carry out the examination
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-09; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients correctly classified by interpreting scintigraphy for the diagnosis of vascular prosthesis infection. The percentage of patients correctly classified is assessed comparing with the diagnostic established by the expert committee. | One year after inclusion when vascular prosthesis infection is suspected and hybrid SPEC-CT with labeled leukocytes has been performed.
  A visual analysis of scintigraphy for diagnosing vascular prosthesis infection. Scintigraphy is considered positive if at least one abnormal localization is seen at vascular prosthesis and if intensity is increasing over time on 20-24h delayed images.

CONTACTS AND LOCATIONS:
Overall Officials: HERVE RAKOTONIRINA, Dr, Principal Investigator — University hospital, Angers, FRANCE
Locations (3):
- France (3):
  - CHU, Angers
  - CH, Le Mans
  - CHRU, Strasbourg